CLINICAL TRIAL: NCT03137888
Title: Pilot Study of Spectroscopic MRI-Guided, Dose-Escalated Radiation Therapy for Newly-Diagnosed Glioblastoma
Brief Title: Spectroscopic MRI-Guided Radiation Therapy Planning in Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Johns Hopkins University (Other); University of Miami (Other); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hui-Kuo Shu, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094188; NCI-2017-00424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD3383-17 (Other: Emory University/Winship Cancer Institute); R01CA214557 (NIH); P30CA138292 (NIH)
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy; Magnetic Resonance Spectroscopy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sMRI-Guided RT with TMZ (Experimental): Patients undergo spectroscopic magnetic resonance imaging-guided dose-escalated radiation therapy daily for the first 5 days of every week (Monday - Friday) over 6 weeks. Patients also receive standard of care temozolomide PO daily during radiation therapy for up to 42 days.
  Interventions: Radiation: Dose-Escalated Radiation Therapy; Procedure: Spectroscopic Magnetic Resonance Imaging; Drug: Temozolomide

INTERVENTIONS:
Radiation: Dose-Escalated Radiation Therapy — Undergo sMRI-guided radiation therapy, dose painted to maximum of 75 Gy over six weeks
  Other Names: RT; Radiation Therapy
Procedure: Spectroscopic Magnetic Resonance Imaging — Patients will undergo sMRI scans within a 14 day window prior to starting treatment
  Other Names: sMRI; MRSI; Magnetic Resonance Spectroscopic Imaging
Drug: Temozolomide — Given PO
  Other Names: Methazolastone; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This pilot clinical trial studies the side effects of spectroscopic magnetic resonance imaging (MRI)-guided radiation therapy and how well it works in treating patients with newly-diagnosed glioblastoma or gliosarcoma. Spectroscopic MRI can show doctors where the extent of tumor is in the brain beyond current clinical MRI scans by mapping areas of high tumor metabolism. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Spectroscopic MRI-guided radiation therapy may work better in treating patients with glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of using spectroscopic MRI (sMRI) to guide dose-escalated radiation therapy (RT) for newly-diagnosed glioblastoma (GBM)s.

II. To determine the safety of using sMRI to guide dose-escalated RT for newly-diagnosed GBMs.

SECONDARY OBJECTIVE:

I. To determine whether the progression free survival at 1 year with sMRI-guided, dose-escalated RT is improved for newly-diagnosed GBMs.

TERTIARY OBJECTIVES:

I. To determine whether sMRI-guided, dose-escalated RT increases the overall survival of patients with newly diagnosed GBMs.

II. To determine whether sMRI data obtained after initiation of therapy (at 2 weeks after RT/TMZ start and prior to cycle 1 and 5 of adjuvant temozolomide [TMZ]) will provide early evidence of GBM progression not seen on standard MRIs.

III. To determine whether performance on neurocognitive and quality-of-life (QOL) assessments in newly-diagnosed GBM patients treated with sMRI-guided, dose-escalated RT differ from historical controls.

OUTLINE:

Patients undergo sMRI-guided radiation therapy daily for the first 5 days of every week (Monday - Friday) over 6 weeks. Patients also receive standard of care temozolomide orally (PO) daily during radiation therapy for up to 42 days.

After completion of study treatment, patients are followed up every 3 months for up to 2 years and then periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a newly-diagnosed glioblastoma or gliosarcoma that has been confirmed pathologically by a board-certified neuropathologist
* Patients must be able to have MRI scans
* Patients must have the following lab values ≤ 14 days prior to registration:

  * White blood cell (WBC) ≥ 3,000/µL
  * Absolute neutrophil count (ANC) ≥ 1,500/µL
  * Platelet count of ≥ 75,000/µL
  * Hemoglobin ≥ 9.0 gm/dL (transfusion is allowed to reach minimum level)
  * Serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2.0 x upper limit of normal (ULN)
  * Bilirubin ≤ 2 x ULN
  * Creatinine ≤ 1.5 mg/dL
* Patients must have a life expectancy of ≥ 12 weeks
* Patients must have a Karnofsky performance status (KPS) ≥ 60
* Patients who are women of childbearing potential must have a negative pregnancy test documented ≤ 14 days prior to registration; this is not specific to dose escalation and is mandatory for standard care for patients being treated with radiation therapy; the cost of this test will be covered by standard of care
* Patients must be able to understand and provide written informed consent
* Members of all races and ethnic groups are eligible for this trial; subjects will be approximately representative of the demographics of the referral base for the participating institutions
* Patient must be able to swallow capsules
* Patients must be willing to forego other cytotoxic and non-cytotoxic therapies against the tumor while being treated on this protocol

Exclusion Criteria:

* Patients with pacemakers, aneurysm clips, neurostimulators, cochlear implants, metal in ocular structures, history of being a steel worker, or other incompatible implants which makes MRI safety an issue are excluded
* Patients that have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy are excluded
* Patients with a history of any other invasive cancer (except non-melanoma skin cancer and excluding carcinoma in-situ), unless in complete remission and off of all therapy for that disease for ≥ 3 years, are ineligible
* Patients with an active infection or serious intercurrent medical illness are ineligible
* Patients receiving any other investigational agents are excluded
* Patients who have received prior cytotoxic, non-cytotoxic or experimental drug therapies for brain tumor are excluded
* Patients with a history of prior cranial radiation are ineligible
* Patients may not be enrolled on any other therapeutic trial for which they are receiving an anti-tumor therapy
* Patients with GBMs located in the following anatomical regions known to have magnetic susceptibility or poor signal will be excluded: mesial temporal lobe, orbitofrontal cortex, prefrontal cortex, medial frontal gyrus, brainstem, and cerebellum
* The maximum radiation target volume for gross tumor volume 3 (GTV3) is 65 cc (per NRG Oncology guide); patient may be excluded after the first sMRI scan if the GTV3 volume is greater than 65 cc (we anticipate that contrast-enhancing tumor volume [residual tumor volume following tumor resection] would be less than 20 cc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Kuo Shu, MD, PhD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trivedi AG, Kim SH, Ramesh KK, Giuffrida AS, Weinberg BD, Mellon EA, Kleinberg LR, Barker PB, Han H, Shu HG, Shim H, Schreibmann E. Applying a Radiation Therapy Volume Analysis Pipeline to Determine the Utility of Spectroscopic MRI-Guided Adaptive Radiation Therapy for Glioblastoma. Tomography. 2023 May 21;9(3):1052-1061. doi: 10.3390/tomography9030086. PMID 37218946
- [Derived] Ramesh K, Gurbani SS, Mellon EA, Huang V, Goryawala M, Barker PB, Kleinberg L, Shu HG, Shim H, Weinberg BD. The Longitudinal Imaging Tracker (BrICS-LIT):A Cloud Platform for Monitoring Treatment Response in Glioblastoma Patients. Tomography. 2020 Jun;6(2):93-100. doi: 10.18383/j.tom.2020.00001. PMID 32548285
- [Derived] Gurbani S, Weinberg B, Cooper L, Mellon E, Schreibmann E, Sheriff S, Maudsley A, Goryawala M, Shu HK, Shim H. The Brain Imaging Collaboration Suite (BrICS): A Cloud Platform for Integrating Whole-Brain Spectroscopic MRI into the Radiation Therapy Planning Workflow. Tomography. 2019 Mar;5(1):184-191. doi: 10.18383/j.tom.2018.00028. PMID 30854456

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | sMRI-Guided RT With TMZ
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | sMRI-Guided RT With TMZ
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: Years] | 56.4 [20.8 to 71.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Successful Co-registration of sMRI-based Treatment Volumes With Clinical Images Into the Radiation Treatment Execution Platform
Description: Feasibility of this approach will be determined by whether treatment volumes based on sMRI can be co-registered with clinical images and transferred into the radiation treatment execution platform in a seamless manner, so that sMRI information can be efficiently applied to the patient treatment.
Time Frame: Up to 2 years after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | sMRI-Guided RT With TMZ
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Incidence of Adverse Event Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: The safety of sMRI to guide dose-escalated RT will be confirmed by assessing toxicity potentially attributable to the RT.
Time Frame: Up to 2 years after completion of therapy
Measure: Number (95% Confidence Interval); unit: Adverse Events
Arm/Group | sMRI-Guided RT With TMZ
Number analyzed (Participants) | 30
Adverse Events | 79 [62 to 99]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Patients were followed at least every 3 months for 2 years from the start of RT.
Time Frame: 2 years from the start of RT.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | sMRI-Guided RT With TMZ
Number analyzed (Participants) | 30
Months | 16.6 [11.6 to 24.0]

4. Other Pre Specified Outcome: Overall Survival (OS)
Description: Patients were followed at least every 3 months for 2.5 years from the start of RT.
Time Frame: 2.5 years from start of RT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | sMRI-Guided RT With TMZ
Number analyzed (Participants) | 30
Months | 23 [18.6 to 27.3]

ADVERSE EVENTS:
Time Frame: Up to 2 years after completion of therapy
Arm/Group | sMRI-Guided RT With TMZ
All-Cause Mortality (participants affected / at risk) | 16/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | sMRI-Guided RT With TMZ (N=30)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Immune system disorders) | 1 (1)
Transaminitis (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Leg edema (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | sMRI-Guided RT With TMZ (N=30)
Abdominal Pain (Gastrointestinal disorders) | 4 (6)
Agitation (Psychiatric disorders) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14)
Anemia (Blood and lymphatic system disorders) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 12 (15)
Anxiety (Psychiatric disorders) | 8 (11)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 12 (16)
Chills (General disorders) | 2 (3)
Cognitive disturbance (Nervous system disorders) | 5 (5)
Concentration Impairment (Nervous system disorders) | 4 (6)
Confusion (Psychiatric disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 16 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Creatinine increased (Investigations) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 8 (13)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dizziness (Nervous system disorders) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema face (General disorders) | 4 (5)
Edema limbs (General disorders) | 5 (5)
Endocrine disorders (Endocrine disorders) | 4 (7)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Erythroderma (Skin and subcutaneous tissue disorders) | 3 (4)
Eye disorders (Eye disorders) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Fatigue (General disorders) | 28 (48)
Fever (General disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 2 (4)
Floaters (Eye disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Gait disturbance (General disorders) | 4 (4)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (5)
General disorders and administration site conditions (General disorders) | 19 (33)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Headache (Nervous system disorders) | 14 (24)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypertension (Vascular disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5)
Infections and infestations (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (9)
Investigations (Investigations) | 2 (7)
Irritability (Psychiatric disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Memory impairment (Nervous system disorders) | 4 (8)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness right-sided (Nervous system disorders) | 2 (2)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 8 (12)
Nausea (Gastrointestinal disorders) | 11 (24)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Nervous system disorders (Nervous system disorders) | 13 (29)
Pain (General disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Paresthesia (Nervous system disorders) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Personality change (Psychiatric disorders) | 2 (3)
Platelet count decreased (Investigations) | 4 (13)
Psychiatric disorders (Psychiatric disorders) | 3 (6)
Renal and urinary disorders (Renal and urinary disorders) | 6 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizure (Nervous system disorders) | 15 (18)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 10 (16)
Thromboembolic event (Vascular disorders) | 3 (3)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (8)
Weight gain (Investigations) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03137888/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03137888/ICF_001.pdf